CLINICAL TRIAL: NCT01401569
Title: STOB-ACTIV: The Efficacy of Exercise and Counseling for Depressed Patients as an Aid for Smoking Cessation, a Randomized Controlled Trial
Brief Title: Efficacy of Exercise and Counseling Intervention on Relapse in Smoker With Depressive Disorders
Acronym: STOB-ACTIV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties for recruiting patients
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8608; n°ID RCB 2010-A00119-30 (Other: Afssaps - French Health Products Safety Agency)
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation; Depression
Keywords: Exercise,; counseling,; smoking cessation,; depressive disorders
MeSH Terms: conditions — Smoking Cessation; Depression; Motor Activity; Depressive Disorder | interventions — Exercise; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): All subjects (intervention and control groups) participate in a smoking cessation program composed of a pharmacological treatment (including nicotine replacement therapy or varenicline) and counseling.
  Interventions: Behavioral: Exercise and counseling (for smoking cessation and physical activity)
- physical activity program (Experimental): Experimental group subjects were required to attend 2 supervised exercise sessions and 2 counseling sessions during Week 1 and Week 2. Supervised exercise and counseling sessions are realized successively. For Week 3 to 8, participants were required to attend 1 supervised exercise session and 1 counseling session plus 1 home exercise session.
  Interventions: Behavioral: Exercise and counseling (for smoking cessation and physical activity)

INTERVENTIONS:
Behavioral: Exercise and counseling (for smoking cessation and physical activity) — Exercise and counseling (for smoking cessation and physical activity)

SUMMARY:
This study investigated the efficacy of an exercise and counseling intervention for depressed smokers (depression subscale of the Hospital Anxiety and Depression Scale, HADS-D score ≥ 8) in term of likelihood of smoking abstinence. Participants were randomized to 8 weeks of intervention: individually delivered exercise and counseling (for smoking cessation and physical activity) or control: health education contact control condition.

DETAILED DESCRIPTION:
This study investigated the efficacy of an exercise and counseling intervention for depressed smokers (depression subscale of the Hospital Anxiety and Depression Scale, HADS-D score ≥ 8) in term of likelihood of smoking abstinence. Participants were randomized to 8 weeks of group delivered exercise and counseling (for smoking cessation and physical activity) or a health education contact control condition. The investigators assess this intervention in a randomized controlled trial of 96 depressed adults smokers recruited by advertisements in local print allocated into one of the two groups (intervention group vs. control group) during a 8-week period and 3 follow-up visits (12, 24, 52 weeks after baseline). All subjects (intervention and control groups) participate in a smoking cessation program composed of a pharmacological treatment (including nicotine replacement therapy or varenicline) and counseling.Experimental group subjects were required to attend 2 supervised exercise sessions and 2 counseling sessions during Week 1 and Week 2. Supervised exercise and counseling sessions are realized successively. For Week 3 to 8, participants were required to attend 1 supervised exercise session and 1 counseling session plus 1 home exercise session.Supervized exercise session consist of 5-min warm-up, 30 min of aerobic activity (stationary bikes), and a 5-min cooldown with stretching. The training intensity is of 60 to 80% maximum heart rate. The sessions are supervised by an exercise specialist who verified and documented the heart rates. Home exercise session consist of 45 min of aerobic exercise (walking, cycling, or running). The training intensity is 6 to 7 on breathlessness visual analog scale.The smoking counseling sessions included the following components: review of a participant's smoking history and motivation to quit, help in the identification of high-risk situations, management of cigarette craving and the generation of problem-solving strategies to deal with such situations.Exercise counseling sessions designed to motivate increased regular physical activity and short bouts of exercise in response to negative affect and urges to smoke. The goal of this intervention was to increase activity level.Health education group subjects were required to participate 75-minute supervised sessions with the same frequency of experimental group. Participants in the health education condition received information on a variety of health topics including sleep hygiene, nutrition, stress and health screening tests for cancer prevention. Participants were also asked to read handouts on health education topics covered during the session.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65 years
* Must be able to give informed consent
* Must live in the area for the next 3 months
* Depression subscale of the Hospital Anxiety and Depression Scale, HADS-D score ≥ 8
* Fagerstrom score > 3
* Must be sedentary, have not participated regularly in aerobic physical exercise (for at least 20 minutes per day, 3 days per week) for the past six months.
* Must be able to exercise at 60% maximum heart rate (MHR) (cleared by a physician)

Exclusion Criteria:

* Cannot read or write fluently in the French language
* Pregnancy or plans to attempt pregnancy
* 60 minutes or more per week of moderate or vigorous physical activity
* Currently in a quit smoking program
* Currently using NRT of any kind or using any other quit smoking method or treatment
* Poor willingness or inability to comply with protocol requirements

Medical problems:

* Cancer treatment within the past 6 monthsPsychiatric Problems
* Currently suicidal or psychotic, (or suicidal/psychotic in last 6 months)
* Taking these specific medications for psychiatric problems: Mood stabilizer (Lithium, Depakote, Neurontin), Antipsychotics (Haldol, Clozaril, Risperdal)
* Currently diagnosis of a bipolar disorder as assessed by MINI 5.0
* Currently diagnosis of a alcohol dependence as assessed by MINI 5.0

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of smoking cessation verified by expired air carbon monoxide | 12 weeks after baseline
  To evaluate whether adding an established exercise and counseling intervention for depressed smokers to a standard smoking cessation treatment program improves smoking outcomes to 12 weeks after baseline ( 7-day point prevalence smoking abstinence verified by expired air carbon monoxide).

SECONDARY OUTCOMES:
prevalence smoking abstinence | (Baseline, 8, 12, 24, 52 weeks after baseline)
  7-day point prevalence smoking abstinence verified by expired air carbon monoxide
Evaluation of Anxiety and Depression | Baseline; 8, 12, 24, 52 weeks after baseline
  The Anxiety and Depression are evaluated by the specific Scale (HADS)
Physical Fitness/Activity | Baseline, 8 weeks 12, 24, 52 weeks after baseline
  Physical Fitness/Activity are evaluated by the 6 minutes Walk Test or TDM6 (Time Frame: Baseline; 8weeks after baseline), by Accelerometry (Time Frame: Baseline; -1, 9 weeks), by the evaluation of Physical self esteem (Time Frame: Baseline; 8, 12 weeks after baseline)with a self-questionnaire (IPAQ7)
Evaluation of Weight | Baseline; 8,12, 24, 52 weeks after baseline
Evaluation of quality of life | Baseline; 8, 12 weeks after baseline
  The quality of life is evaluated by a self-questionnaire (SF-12)
Cigarette Craving | Baseline; 8, 12 weeks after baseline
  The Cigarette Craving is evaluated by self-questionnaires: QSU and Fagerström test
Smoking Abstinence self Efficacy | Baseline; 8, 12 weeks after baseline
  The Smoking Abstinence self Efficacy is evaluated by the self-questionnaire (CSQ 12)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Bernard P, Ninot G, Cyprien F, Courtet P, Guillaume S, Georgescu V, Picot MC, Taylor A, Quantin X. Exercise and Counseling for Smoking Cessation in Smokers With Depressive Symptoms: A Randomized Controlled Pilot Trial. J Dual Diagn. 2015;11(3-4):205-16. doi: 10.1080/15504263.2015.1113842. PMID 26683252